CLINICAL TRIAL: NCT05153083
Title: Cryoablation of Intercostal Nerves for Better Control of Postoperative Pain After Thoracic and Thoracoabdominal Open Surgery - A Physician-initiated, International, Multicentre, Prospective, Observational Registry of Patients Undergoing Open Thoracic (TAA) and Thoracoabdominal Aortic Aneurysms Repair (TAAA) Using Cryoablation of Intercostal Nerves to Improve Postoperative Pain Control. (Cryo Registry)
Brief Title: Cryoablation of Intercostal Nerves for Better Control of Postoperative Pain After Thoracic and Thoracoabdominal Open Surgery
Status: Suspended | Type: Observational
Why Stopped: unavailability of cryoablation probes
Sponsor: Germano Melissano (Other)
Responsible Party: Sponsor-Investigator, Germano Melissano, Prof, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: Cryo Registry
Record Dates: First submitted 2021-11-19; First posted 2021-12-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient undergoing open thoracic (TAA) and thoracoabdominal aortic aneurysms repair (TAAA): Subjects undergoing open thoracic (TAA) and thoracoabdominal aortic aneurysms repair (TAAA) using cryoablation of intercostal nerves
  Interventions: Procedure: Open thoracic (TAA) and thoracoabdominal aortic aneurysms repair (TAAA)

INTERVENTIONS:
Procedure: Open thoracic (TAA) and thoracoabdominal aortic aneurysms repair (TAAA) — Each participating center will be able to use its preferred European Conformity marked device, for cryoablation according to their normal clinical practice and according to the instructions for use.

SUMMARY:
The purpose of the registry is to evaluate the peri-operative and short- term outcomes of intercostal nerves cryoablation for post-operative pain control after open thoracic and thoracoabdominal aortic aneurysms repair.

The cryoablation procedure is one of the opportunities for pain control after thoracotomy. So, it is routinely performed in major several centers in aortic surgery around the world as a part of the TAA and TAAA procedure.

The Registry will include approximately 200 patients treated from January 2022 to January 2024 for thoracic or thoracoabdominal aortic aneurysm by means of open surgery and in whom intraoperative intercostal nerves cryoablation will be performed; to reach 200 patients, the enrolments can be extended until January 2027.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years
* Patients who will undergo TAA and TAAA open repair with intraoperative intercostal nerves cryoablation
* Subject has consented for study participation and signed the approved Informed Consent

Exclusion Criteria:

* Patients with active systemic or cutaneous infection or inflammation
* Patients who are pregnant or breastfeeding
* Patients younger than 18 years of age
* Unwilling or unable to comply with the follow-up schedule
* Inability or refusal to give informed consent
* Frank rupture
* Previous stroke with neurological sequelae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Registry will include approximately 200 patients treated from January 2022 to January 2024 for thoracic or thoracoabdominal aortic aneurysm by means of open surgery and in whom intraoperative intercostal nerves cryoablation will be performed; .
  to reach 200 patients, the enrolments can be extended until January 2027.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
technical success | From Admission to 1 years
  Freedom from Death
change in dose of narcotic administration | From Admission to 1 years
  reduction opioids usage for thoracic incision pain
Primary clinical success | up to 3 weeks
  pain control defined as a visual analogic scale < 5 in the perioperative period up to the discharge
secondary clinical success | up to 3 weeks
  pain control in in the perioperative period up to the discharge, using analgesic non opioids drugs

CONTACTS AND LOCATIONS:
Locations (13):
- Hospital Hietzing,Vienna, Vienna, Austria
- Salpetriere University Hospital, Paris, France
- Germany (5):
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - University Medical Center Hamburg, Hamburg
  - Hannover Medical School, Hanover
  - Saarland University Hospital, Homburg
- Italy (2):
  - Policlinico S. Orsola - Malpighi, Bologna, Italy
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy
- Maastricht University Medical Center, Maastricht, Netherlands
- Centro Hospitalar de Entre o Douro e Vouga, Santa Maria da Feira, Portugal
- University Hospital of Bern, Bern, Switzerland
- St Bartholomew's Hospital, London, United Kingdom

REFERENCES:
- [Background] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735
- [Background] Richardson J, Sabanathan S, Shah R. Post-thoracotomy spirometric lung function: the effect of analgesia. A review. J Cardiovasc Surg (Torino). 1999 Jun;40(3):445-56. PMID 10412938
- [Background] Carlsson CA, Persson K, Pelletieri L. Painful scars after thoracic and abdominal surgery. Acta Chir Scand. 1985;151(4):309-11. PMID 4036485
- [Background] Soto RG, Fu ES. Acute pain management for patients undergoing thoracotomy. Ann Thorac Surg. 2003 Apr;75(4):1349-57. doi: 10.1016/s0003-4975(02)04647-7. PMID 12683601
- [Background] Gottschalk A, Cohen SP, Yang S, Ochroch EA. Preventing and treating pain after thoracic surgery. Anesthesiology. 2006 Mar;104(3):594-600. doi: 10.1097/00000542-200603000-00027. No abstract available. PMID 16508407
- [Background] Clemence J Jr, Malik A, Farhat L, Wu X, Kim KM, Patel H, Yang B. Cryoablation of Intercostal Nerves Decreased Narcotic Usage After Thoracic or Thoracoabdominal Aortic Aneurysm Repair. Semin Thorac Cardiovasc Surg. 2020 Autumn;32(3):404-412. doi: 10.1053/j.semtcvs.2020.01.008. Epub 2020 Jan 20. PMID 31972300
- [Background] Johnston KW, Rutherford RB, Tilson MD, Shah DM, Hollier L, Stanley JC. Suggested standards for reporting on arterial aneurysms. Subcommittee on Reporting Standards for Arterial Aneurysms, Ad Hoc Committee on Reporting Standards, Society for Vascular Surgery and North American Chapter, International Society for Cardiovascular Surgery. J Vasc Surg. 1991 Mar;13(3):452-8. doi: 10.1067/mva.1991.26737. PMID 1999868
- [Background] Chaikof EL, Fillinger MF, Matsumura JS, Rutherford RB, White GH, Blankensteijn JD, Bernhard VM, Harris PL, Kent KC, May J, Veith FJ, Zarins CK. Identifying and grading factors that modify the outcome of endovascular aortic aneurysm repair. J Vasc Surg. 2002 May;35(5):1061-6. doi: 10.1067/mva.2002.123991. No abstract available. PMID 12021728
- [Background] Achouh PE, Madsen K, Miller CC 3rd, Estrera AL, Azizzadeh A, Dhareshwar J, Porat E, Safi HJ. Gastrointestinal complications after descending thoracic and thoracoabdominal aortic repairs: a 14-year experience. J Vasc Surg. 2006 Sep;44(3):442-6. doi: 10.1016/j.jvs.2006.05.018. PMID 16950413
- [Background] Riambau V, Bockler D, Brunkwall J, Cao P, Chiesa R, Coppi G, Czerny M, Fraedrich G, Haulon S, Jacobs MJ, Lachat ML, Moll FL, Setacci C, Taylor PR, Thompson M, Trimarchi S, Verhagen HJ, Verhoeven EL, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus ES, Hinchliffe RJ, Kakkos S, Koncar I, Lindholt JS, Vega de Ceniga M, Vermassen F, Verzini F, Document Reviewers, Kolh P, Black JH 3rd, Busund R, Bjorck M, Dake M, Dick F, Eggebrecht H, Evangelista A, Grabenwoger M, Milner R, Naylor AR, Ricco JB, Rousseau H, Schmidli J. Editor's Choice - Management of Descending Thoracic Aorta Diseases: Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2017 Jan;53(1):4-52. doi: 10.1016/j.ejvs.2016.06.005. No abstract available. PMID 28081802